CLINICAL TRIAL: NCT00059579
Title: Functional MRI Study of Brain Mechanism Mediating Anhedonia in Major Depression
Brief Title: Brain Regulation of Emotions in People With Depression and Anhedonia
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030149; 03-M-0149
Record Dates: First submitted 2003-04-29; First posted 2003-04-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-12

CONDITIONS: Major Depressive Disorder
Keywords: Reward; Cortex; Dopamine; Neuroimaging; Strirtum; Major Depressive Disorder (MDD); Melancholic Features; Brain Imaging; Functional Magnetic Resonance Imaging (fMRI); Dopaminergic Mechanisms; Anhedonia; Depression; Major Depressive Disorder; MDD; Healthy Volunteer; HV
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia; Depression

SUMMARY:
This study will use magnetic resonance imaging (MRI) to examine how the brain regulates emotions in healthy people and in patients who have major depression and anhedonia (loss of feeling of pleasure in things that normally give pleasure).

Healthy normal volunteers and patients between 18 and 50 years of age with major depression, with or without significant anhedonia, are eligible for this study. Candidates will be screened with a psychiatric interview, a physical examination that will include blood and urine samples, and an electrocardiogram, and a questionnaire about their emotions.

Participants will perform a monetary reward task while lying in an MRI scanner. The task is similar to playing a computer video game with the possibility of winning cash. The amount of cash is largely dependent on the subject's performance. The accumulated amount of cash earned in a session will fluctuate depending on the subject's continuing performance level. That is, during a single session, a subject could lose money earned early in the session if his or her performance later in the session is not as good as earlier.

MRI pictures will be taken during performance of the task. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The patient lies on a table that is moved into the scanner (a narrow cylinder) and wears earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure will last about 1 to 1-1/2 hours.

DETAILED DESCRIPTION:
Anhedonia has been one of the two key diagnostic criteria for major depressive disorder (MDD) since the publication of The Diagnostic and Statistical Manual of Mental Disorders, Third Edition, yet little is known about its neural substrates. Neuroimaging studies have identified numerous brain regions that are thought to be involved with MDD. Most studies dealt with MDD as a syndromal entity, and not surprisingly, yielded quite variable results with respect to the areas of the brain identified, the nature of the functional changes (i.e., decrease or increase in activities), lateralization, and correlation with clinical symptoms. Clinical heterogeneity and lack of symptom-specific targets are presumably among the factors contributing to the variability. The hypothesis that a functionally impaired mesolimbic dopaminergic pathway may comprise a part of neural substrate underlying core MDD symptoms of anhedonia and loss of motivation has been proposed. Nevertheless, the roles of brain reward mechanisms in mediating anhedonia in MDD remain unclear. Availability of appropriate experimental paradigms that can be used empirically to measure anhedonia is a prerequisite to test such a hypothesis. Recent studies using monetary incentive paradigms coupled with neuroimaging techniques have identified hemodynamic responses in structures that serve as part of the mesolimbic dopaminergic pathway during processing rewards in healthy humans.

We hypothesize that anhedonia in MDD is associated with impairment of brain reward mechanisms such that dysfunction of the orbital and ventromedial frontal cortices involved in the impaired hedonic attribution capacity, while dysfunction of the ventral striatum area that contains the nucleus accumbens is involved with the reduced or lack of reactivity to rewarding environmental stimuli in patients with MDD. Our hypothesis is to link specific neural substrates to the two psychiatric components of anhedonia, i.e., loss of interest and lack of reactivity, as defined in the diagnostic criteria for MDD. We plan to operationally test our hypothesis by using empirical measurement of reward responses in MDD patients with and without significant anhedonia using a conditioning task assessing appetitive and aversive learning without any performance aspects and spatial delayed response task assessing the relationship between reward, performance and mood with the event-related functional magnetic resonance imaging method. We expect to find reduced activation of the ventral striatum, orbital and ventromedial frontal cortices in response to monetary incentive stimuli in MDD patients with significant anhedonia relative to MDD patients without anhedonia and healthy control.

In order to assess the role of dopamine in anhedonia and in reward processing, we propose to assess the effect of dietary tyrosine plus phenylalanine depletion on the neural and behavioral responses associated with the performing of the monetary reward tasks investigated herein in an additional sample of subjects. Dietary depletion of tyrosine and phenylalanine, two DA precursors, is a validated method to induce significant reduction of the brain DA concentration as shown in two previous [11C]Raclopride PET studies. We hypothesize that depressed patients will show less activation than controls in brain regions associated with the mesolimbic DA system, such as striatum, amygdala, anterior cingulate gyrus and orbitofrontal cortex in response to reward in the placebo condition. We expect tyrosine and phenylalanine depletion to induce a similar neural impairment to reward in healthy subjects, including a reduction of the neural activation in the striatum, amygdala, anterior cingulate gyrus and orbitofrontal cortex in response to reward. The reduction of the neural activation in those regions will be stronger in healthy controls than in depressed patients. Finally, we hypothesize that tyrosine depletion will influence negatively the valence ratings of rewarding stimuli in healthy subjects. In depressed patients, anhedonia scores will correlate negatively with the valence ratings of rewarding stimuli in the placebo condition already.

The outcome of the proposed work may provide clues for diagnosis, classification, and treatment of MDD, and may also yield leads for identifying the fundamental neural mechanisms underlying anhedonia in other disabling psychiatric conditions such as schizophrenia and addiction.

ELIGIBILITY:
* INCLUSION CRITERIA

For both patient and control groups:

Age 18 to 50 of any ethnicity without other significant medical conditions

Not in active use of illicit drugs and heavy consumption of alcohol

No metallic implants or onplants that are ferromagnetic

Competent to sign consent forms to participate in the study.

For patient groups:

For the group with significant anhedonia, current MDD, as defined by DSM-IV criteria, with significant anhedonia defined as having PAS and/or SAS scores at or above one standard deviation of appropriate norm. For the group without significant anhedonia, current MDD, as defined by DSM-IV criteria, without significant anhedonia defined as having PAS and/or SAS scores within or below one standard deviation of appropriate norm. The BPD subjects will meet DSM-IV criteria for bipolar I or II disorder, most recent episode depressed and will currently be in a major depressive episode. We will use the Young Mania Rating Scale to assess the severity of the disorder Subjects may be enrolled as either inpatients or outpatients at their entrance to the study.

For control group:

No prior history of any psychiatric conditions including substance dependence

No family history of MDD, bipolar disorder, or psychosis

PAS and/or SAS scores within or below one standard deviation of appropriate norm.

EXCLUSION CRITERIA:

Medical conditions or concomitant medications that are likely to influence cerebral blood flow or neurological function including cardiovascular, respiratory, endocrine and neurological diseases;

History of psychosis, current mania and substance dependence;

Exposure to psychiatric medications in the past 4 weeks;

History of repeated self-mutilation or homicidal attempts, current active suicidal / homicidal ideations;

Current or recent (within past six weeks) illicit drug use or heavy alcohol consumption (more than 2 six-packs of beer or equivalent alcoholic beverages per week);

Pathological gamblers as defined by DSM-IV.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2003-04-24; Study Completion 2010-11-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blanchard JJ, Horan WP, Brown SA. Diagnostic differences in social anhedonia: a longitudinal study of schizophrenia and major depressive disorder. J Abnorm Psychol. 2001 Aug;110(3):363-71. doi: 10.1037//0021-843x.110.3.363. PMID 11502079
- [Background] Boyer P, Tassin JP, Falissart B, Troy S. Sequential improvement of anxiety, depression and anhedonia with sertraline treatment in patients with major depression. J Clin Pharm Ther. 2000 Oct;25(5):363-71. doi: 10.1046/j.1365-2710.2000.00302.x. PMID 11123488
- [Background] Barbier EL, Silva AC, Kim SG, Koretsky AP. Perfusion imaging using dynamic arterial spin labeling (DASL). Magn Reson Med. 2001 Jun;45(6):1021-9. doi: 10.1002/mrm.1136. PMID 11378880